CLINICAL TRIAL: NCT06144099
Title: Prothrombin Complex Concentrate and Fresh Frozen Plasma in Viscoelastic Test-based Goal-directed Bleeding Management in Non-Cardiac Surgery
Brief Title: Prothrombin Complex Concentrate vs Fresh Frozen Plasma in Goal-directed Bleeding Management in Non-cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC22195220002002
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Spine, Open; Hip Osteoarthritis; Knee Disease
MeSH Terms: conditions — Prostatic Neoplasms; Spinal Dysraphism; Osteoarthritis, Hip | interventions — Factor IX

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fresh frozen plasma (Active Comparator): according to the Thromboelastography (TEG) test, CK r-time prolongation, fresh frozen plasma transfusion (FFP) is performed
  Interventions: Biological: fresh frozen plasma
- prothrombin complex concentrate (Experimental): according to the Thromboelastography (TEG) test, CK r-time prolongation,prothrombin complex concentrate (PCC) administration
  Interventions: Biological: prothrombin complex concentrate

INTERVENTIONS:
Biological: fresh frozen plasma — transfusion of fresh frozen plasma
  Arms: fresh frozen plasma
Biological: prothrombin complex concentrate — prothrombin complex concentrate administration
  Arms: prothrombin complex concentrate

SUMMARY:
The primary endpoint of this study is the completion time of hemostasis treatment when administered Fresh frozen plasma (FFP) and frozen powder coagulation factor concentrate (PCC) in goal-directed bleeding management for non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing spine surgery
* patients undergoing open radical prostatectomy
* patients undergoing hip arthroplasty
* patients undergoing knee arthroplasty

Exclusion Criteria:

* Patients taking oral anticoagulants,
* Patient taking recombinant factor VII a
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
duration from the time diagnosing r-time prolongation to the time achieving bleeding control | 1 min

SECONDARY OUTCOMES:
Red Blood Cell amount | 1 hour
  Red Blood Cell transfusion amount during surgery
FFP amount | 1 hour
  FFP transfusion amount during surgery
Platelet amount | 1 hour
  Platelet transfusion amount during surgery
r-time | 10 min
  CK r-time after PCC or FFP
CRT-MA | 10 min
  CRT-MA after PCC or FFP
CFF-MA | 10 min
  CFF-MA after PCC or FFP
Bleeding | 6 hour
  Postoperative bleeding amount
oxygenation profile | 1 hour
  PaO2/FiO2 ratio

IPD SHARING:
Plan to Share IPD: Undecided